CLINICAL TRIAL: NCT00191113
Title: Humatrope Treatment to Final Height in Turner's Syndrome
Brief Title: Somatropin Treatment to Final Height in Turner Syndrome
Acronym: GDCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly and Company
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 817/4419; #817 B9R-CA-GDCT Core study; #4419 GDCT/1 Addenda
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2010-01-27 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2009-12

CONDITIONS: Turner Syndrome
Keywords: syndrome; Turner; Turner's; height; growth; growth hormone; somatropin; short stature; short; hearing; glucose metabolism
MeSH Terms: conditions — Turner Syndrome; Syndrome; Dwarfism | interventions — Human Growth Hormone; Growth Hormone; Ethinyl Estradiol; Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Control arm; untreated with Humatrope. Ethinyl estradiol (escalating doses to 20 mcg daily) after age 13, and medroxyprogesterone acetate (10 mg tablets ten days monthly) after age 15. Subject continues until Core study completion criteria are met (protocol final height).
  Interventions: Drug: Ethinyl estradiol; Drug: Medroxyprogesterone acetate
- Humatrope (Experimental): Humatrope (0.05 mg/kg/dose) by subcutaneous injection 6 times per week. Ethinyl estradiol (escalating doses to 20 mcg daily) after age 13, and medroxyprogesterone acetate (10 mg tablets ten days monthly) after age 15. Subject continues until Core study completion criteria are met (protocol final height).
  Interventions: Drug: Somatropin; Drug: Ethinyl estradiol; Drug: Medroxyprogesterone acetate

INTERVENTIONS:
Drug: Somatropin — 0.05 mg/kg/dose by subcutaneous injection 6 times per week, until Core study completion criteria are met (protocol final height).
  Other Names: Humatrope; Growth hormone
  Arms: Humatrope
Drug: Ethinyl estradiol — escalating doses 2.5-20.0 mcg tablets daily after age 13 and at least one year on study, continuing until Core study completion criteria are met.
Drug: Medroxyprogesterone acetate — 10 mg tablets, ten days monthly, after age 15, continuing until Core study completion criteria are met.

SUMMARY:
A randomized, controlled trial in girls with Turner syndrome at least 7 years old and younger than 13 at study entry, to determine the efficacy and safety of Humatrope (somatropin) treatment in promoting linear growth to final height.

DETAILED DESCRIPTION:
A randomized, controlled trial of Humatrope (somatropin) treatment in girls with Turner syndrome at least 7 years old and younger than 13 at study entry.

Core study objectives are to determine the efficacy of Humatrope in promoting linear growth to final height in girls with Turner syndrome, and to assess the safety of this treatment. Core study completion criteria (protocol final height) are that the patient has both a height velocity < 2 cm per year and a bone age of 14 years or greater.

Addendum 1 provides the option of Humatrope treatment to patients who were randomized to the Control arm of the Core study and who discontinued from the study on or after December 19, 1997.

Addendum 2 objectives are: 1) to collect true final height data; 2) to evaluate hearing, tympanic membrane function and other specific areas of interest with respect to the safety of growth hormone therapy in Turner syndrome; 3) to evaluate pancreatic beta cell function (glucose metabolism) in patients previously enrolled in the Core study.

Addendum 3 objective is to determine the parental origin of the retained X chromosome of an appropriate subset of patients currently or previously enrolled in the Core study, and to determine whether this parental origin holds any predictive value for spontaneous growth or for response to growth hormone therapy.

ELIGIBILITY:
Inclusion Criteria:

* girl with Turner syndrome
* prepubertal, Tanner stage I breast
* height velocity less than 6 cm/year and height less than or equal to the tenth percentile for sex and age in general population
* at least 6 months (preferably 12 months) of accurate height measurements available for calculation of pre-study height velocity
* if thyroxine deficient, to have received replacement therapy, and for six months prior to enrollment have had normal thyroid function tests

Exclusion Criteria:

* prior treatment with growth hormone
* presence of a Y component in karyotype with gonads in situ
* diabetes mellitus

Ages: 7 Years to 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 1989-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- Canada (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halifax, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingston, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sainte-Foy, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec

REFERENCES:
- [Background] Lyon AJ, Preece MA, Grant DB. Growth curve for girls with Turner syndrome. Arch Dis Child. 1985 Oct;60(10):932-5. doi: 10.1136/adc.60.10.932. PMID 4062345
- [Background] Kuczmarski RJ, Ogden CL, Grummer-Strawn LM, Flegal KM, Guo SS, Wei R, Mei Z, Curtin LR, Roche AF, Johnson CL. CDC growth charts: United States. Adv Data. 2000 Jun 8;(314):1-27. PMID 11183293
- [Result] Hamelin CE, Anglin G, Quigley CA, Deal CL. Genomic imprinting in Turner syndrome: effects on response to growth hormone and on risk of sensorineural hearing loss. J Clin Endocrinol Metab. 2006 Aug;91(8):3002-10. doi: 10.1210/jc.2006-0490. Epub 2006 Jun 6. PMID 16757526
- [Result] Stephure DK; Canadian Growth Hormone Advisory Committee. Impact of growth hormone supplementation on adult height in turner syndrome: results of the Canadian randomized controlled trial. J Clin Endocrinol Metab. 2005 Jun;90(6):3360-6. doi: 10.1210/jc.2004-2187. Epub 2005 Mar 22. PMID 15784709
- [Derived] Taback SP, Van Vliet G. Health-related quality of life of young adults with Turner syndrome following a long-term randomized controlled trial of recombinant human growth hormone. BMC Pediatr. 2011 May 29;11:49. doi: 10.1186/1471-2431-11-49. PMID 21619701
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Addenda 1, 2, and 3 are not sequential, and they differ in eligibility criteria. Depending on individual eligibility and choices made, a patient might have participated in none, 1, 2, or all 3 of these addenda.
Pre-assignment Details: Addendum 1: provided option of Humatrope treatment to patients who had been randomized to control in Core Study. Addendum 2: extended period of follow-up for 5 years after discontinuation from Core Study. Addendum 3: evaluated possible genomic imprinting effects (published: Hamelin et al. 2006).
Groups:
- As-Randomized Control: Control arm; untreated with Humatrope. Ethinyl estradiol (escalating doses to 20 mcg daily) after age 13, and medroxyprogesterone acetate (10 mg tablets ten days monthly) after age 15. Subject continues until Core study completion criteria are met (protocol final height).
- As-Randomized Humatrope: Humatrope (0.05 mg/kg/dose) by subcutaneous injection 6 times per week. Ethinyl estradiol (escalating doses to 20 mcg daily) after age 13, and medroxyprogesterone acetate (10 mg tablets ten days monthly) after age 15. Subject continues until Core study completion criteria are met (protocol final height).
Period: Core Study
Arm/Group | As-Randomized Control | As-Randomized Humatrope
Started | 78 | 76
Completed | 43 | 61
Not Completed | 35 | 15
Not completed — Withdrawal by Subject | 25 | 9
Not completed — Protocol Violation | 6 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Death | 1 | 0
Period: Addendum 1
Arm/Group | As-Randomized Control | As-Randomized Humatrope
Started | 2 | 0 (Not Applicable -- only Control patients were eligible for Addendum 1)
Completed | 2 | 0 (Not Applicable -- only Control patients were eligible for Addendum 1)
Not Completed | 0 | 0
Period: Addendum 2
Arm/Group | As-Randomized Control | As-Randomized Humatrope
Started | 28 | 48
Completed | 18 | 31
Not Completed | 10 | 17
Period: Addendum 3
Arm/Group | As-Randomized Control | As-Randomized Humatrope
Started | 20 | 37
Completed | 20 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | As-Randomized Control | As-Randomized Humatrope | Total
Number analyzed (Participants) | 78 | 76 | 154
Age Continuous [Mean (Standard Deviation); unit: years] | 10.46 (1.77) | 10.36 (1.80) | 10.41 (1.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 76 | 154
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 78 | 76 | 154
Karyotype [Number; unit: participants]
  45,X | 48 | 45 | 93
  45,X/46,XXqi | 6 | 2 | 8
  45,X/46,XXr | 1 | 2 | 3
  45,X/46,XX | 3 | 3 | 6
  46,XXqi | 2 | 6 | 8
  45,X/47,XXX | 1 | 2 | 3
  46,XXp | 1 | 0 | 1
  45,X/46,XXp | 1 | 1 | 2
  45,X/46,XX/47,XXX | 0 | 0 | 0
  46,XXr | 0 | 0 | 0
  Other | 15 | 15 | 30
Race/Ethnicity [Number; unit: participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 7 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 54 | 66 | 120
  Hispanic | 0 | 2 | 2
  Other | 4 | 0 | 4
  Unknown | 11 | 1 | 12
Bone Age [Mean (Standard Deviation); unit: years] — Bone age was determined by the Greulich-Pyle method.
  years | 8.57 (1.51) | 8.79 (1.42) | 8.69 (1.46)
Height [Mean (Standard Deviation); unit: centimeters] | 120.06 (8.26) | 119.84 (8.45) | 119.96 (8.33)
Height Standard Deviation Score (SDS) [Lyon] [Mean (Standard Deviation); unit: Standard Deviation Score (SDS)] — SDS report the number of standard deviations from the mean for age and sex for an individual measurement (normal range: -2 to +2 SDS). Height SDS [Lyon] uses the Turner syndrome reference height values for age (Lyon AJ et al. 1985) as the population mean and standard deviation. Height SDS is derived by subtracting the population mean from individual's height value and then dividing that difference by the population standard deviation. Since the data reported by Lyon AJ et al represent a Turner syndrome reference standard, values for patients with Turner syndrome are centered around zero.
  Standard Deviation Score (SDS) | -0.13 (0.86) | -0.10 (0.88) | -0.11 (0.87)
Height Standard Deviation Score (SDS) [National Center for Health Statistics (NCHS)] [Mean (Standard Deviation); unit: Standard Deviation Score (SDS)] — SDS report the number of standard deviations from the mean for age and sex for an individual measurement (normal range: -2 to +2 SDS). Height SDS [NCHS] uses the NCHS US general female population reference height values for age (Kuczmarski RJ et al. 2000) as the population mean and standard deviation. Calculation of Height SDS is provided in Height SDS [Lyon] description (baseline). Since data reported by Kuczmarski RJ et al provides US general female population standards, values of Height SDS [NCHS] for untreated patients with Turner syndrome tend to be below zero e.g, -2.0 to -4.0 SDS.
  Standard Deviation Score (SDS) | -3.25 (0.82) | -3.21 (0.82) | -3.23 (0.82)

OUTCOME MEASURES:

1. Primary Outcome: Height Standard Deviation Score (SDS) (National Center for Health Statistics [NCHS]), Change From Baseline to Last Measurement, As Randomized Population
Description: Value analyzed is change from baseline to the most mature height measurement available. The terms Standard Deviation Score (SDS) and National Center for Health Statistics (NCHS) were defined in baseline characteristics. Greater height SDS values indicate greater height; positive values of change from baseline indicate increased height.
Time Frame: Baseline, and end of 4-year addendum
Population: Population of all randomized patients. Intent to treat analysis with as-randomized treatment groups, at most mature measurement available.
Measure: Least Squares Mean (Standard Error); unit: Standard Deviation Score (SDS) [NCHS]
Arm/Group | As-Randomized Control | As-Randomized Humatrope
Number analyzed (Participants) | 78 | 76
Standard Deviation Score (SDS) [NCHS] | 0.09 (0.07) | 0.97 (0.07)
Statistical Analysis 1: Comparison: As-Randomized Control vs As-Randomized Humatrope; This component of the primary analysis is inferential i.e. to ascertain definitively whether Humatrope treatment affects change in Height SDS (NCHS). Null hypothesis is no effect of Humatrope treatment; Test type: Superiority or Other; p < 0.001, ANCOVA; Model includes baseline height SDS, baseline age, treatment, and interactions. Age and interaction terms removed when not significant; Mean Difference (Final Values) = 0.9, 95% CI [0.7 to 1.1] — Effect direction is "As-Randomized Humatrope" minus "As-Randomized Control"

2. Primary Outcome: Height Standard Deviation Score (SDS) (National Center for Health Statistics [NCHS]), Last Measurement After Attainment of Final Height
Description: SDS report the number of standard deviations from the mean for age and sex for an individual measurement (normal range: -2 to +2 SDS). Height SDS [NCHS] uses the NCHS US general female population reference height values for age (Kuczmarski RJ et al. 2000) as the population mean and standard deviation. Calculation of Height SDS is provided in Height SDS [Lyon] description (Baseline). Since data reported by Kuczmarski RJ et al provides US general female population standards, values of Height SDS [NCHS] for untreated patients with Turner syndrome tend to be below zero e.g, -2.0 to -4.0 SDS.
Time Frame: at completion of core study, or at end of 4-year addendum
Population: Population of patients for whom Final Height measurements are available. Efficacy analysis with as-treated treatment groups, at most mature measurement available at or after attainment of Final Height.
Measure: Least Squares Mean (Standard Error); unit: Standard Deviation Score (SDS) [NCHS]
Groups:
- As-Treated No Growth Hormone: Patients who never received growth hormone
- As-Treated Growth Hormone: Patients who received Humatrope or another brand of growth hormone
Arm/Group | As-Treated No Growth Hormone | As-Treated Growth Hormone
Number analyzed (Participants) | 48 | 82
Standard Deviation Score (SDS) [NCHS] | -3.30 (0.07) | -2.25 (0.05)
Statistical Analysis 1: Comparison: As-Treated No Growth Hormone vs As-Treated Growth Hormone; Estimation analysis of the magnitude of effect of treatment with growth hormone upon Final Height. Null hypothesis is no effect of growth hormone upon attained height standard deviation score (National Center for Health Statistics); Test type: Superiority or Other; p < 0.001, ANCOVA; Model includes baseline height SDS, baseline age, treatment, and interactions. Age and interactions terms removed when not significant; Mean Difference (Final Values) = 1.0, 95% CI [0.9 to 1.2] — Effect direction is "As-Treated Growth Hormone" minus "As-Treated No Growth Hormone"

3. Secondary Outcome: Height Standard Deviation Score (SDS) (National Center for Health Statistics [NCHS]), Change From Baseline, As-Treated Population
Description: as for outcome 1
Time Frame: every 3 months during core study, and at start and end of 4-year addendum
Measure: Least Squares Mean (Standard Error); unit: Standard Deviation Score (SDS) [NCHS]
Groups:
- As-Treated Growth Humatrope: Patients who received Humatrope or another brand of growth hormone
Arm/Group | As-Treated No Growth Hormone | As-Treated Growth Humatrope
Number analyzed (Participants) | 48 | 82
Standard Deviation Score (SDS) [NCHS] | -0.09 (0.08) | 0.99 (0.06)
Statistical Analysis 1: Comparison: As-Treated No Growth Hormone vs As-Treated Growth Humatrope; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 1.1, 95% CI [0.9 to 1.3]

4. Secondary Outcome: Height (Centimeters [cm])
Description: Most mature measurement available, at or after attainment of Final Height.
Time Frame: every 3 months during core study, and at start and end of 4-year addendum
Measure: Least Squares Mean (Standard Error); unit: centimeters (cm)
Arm/Group | As-Treated No Growth Hormone | As-Treated Growth Humatrope
Number analyzed (Participants) | 48 | 82
centimeters (cm) | 141.63 (0.47) | 148.52 (0.36)
Statistical Analysis 1: Comparison: As-Treated No Growth Hormone vs As-Treated Growth Humatrope; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 6.9, 95% CI [5.7 to 8.1]

5. Secondary Outcome: Number of Participants With an Abnormal Pure Tone Audiometry, Audiologist Assessment
Time Frame: at completion of core study or beginning of addendum
Population: All Randomized Patients with Hearing Examination
Measure: Number; unit: participants
Arm/Group | As-Treated No Growth Hormone | As-Treated Growth Hormone
Number analyzed (Participants) | 19 | 53
participants | 10 | 29
Statistical Analysis 1: Comparison: As-Treated No Growth Hormone vs As-Treated Growth Hormone; Test type: Superiority or Other; p > 0.999, Fisher Exact

6. Secondary Outcome: Number of Participants With Abnormal Speech Audiometry, Audiologist Assessment
Time Frame: at completion of core study or beginning of addendum
Population: All Randomized Patients with Hearing Examination
Measure: Number; unit: participants
Arm/Group | As-Treated No Growth Hormone | As-Treated Growth Hormone
Number analyzed (Participants) | 19 | 53
participants | 3 | 12
Statistical Analysis 1: Comparison: As-Treated No Growth Hormone vs As-Treated Growth Hormone; Test type: Superiority or Other; p = 0.744, Fisher Exact

7. Secondary Outcome: Number of Participants With Abnormal Impedance Tympanometry, Audiologist Assessment
Time Frame: at completion of core study or beginning of addendum
Population: All Randomized Patients with Hearing Examination
Measure: Number; unit: participants
Arm/Group | As-Treated No Growth Hormone | As-Treated Growth Hormone
Number analyzed (Participants) | 19 | 53
participants | 2 | 18
Statistical Analysis 1: Comparison: As-Treated No Growth Hormone vs As-Treated Growth Hormone; Test type: Superiority or Other; p = 0.073, Fisher Exact

8. Secondary Outcome: Number of Participants With Hearing Loss, Audiologist Assessment
Description: Sensorineural Hearing Loss (SNHL)=air conduction threshold >20 dB HL and air-bone gap ≤10 dB HL; Conductive Hearing Loss (CHL)= air conduction threshold >20 dB HL, bone conduction threshold ≤20 dB HL and air-bone gap >10 dB HL; Mixed Hearing Loss (MHL) = evidence of SNHL as defined above and CHL as defined above, in the same ear; Unspecified Hearing Loss (UHL)= abnormal hearing with none of SNHL, CHL, or MHL present.
Time Frame: at completion of core study or beginning of addendum
Population: All Randomized Patients with Hearing Examination for whom Audiologist responded to Hearing Loss question
Measure: Number; unit: participants
Arm/Group | As-Treated No Growth Hormone | As-Treated Growth Hormone
Number analyzed (Participants) | 19 | 52
participants
  Conductive Hearing Loss | 1 | 7
  Sensorineural Hearing Loss | 8 | 15
  Mixed Hearing Loss | 2 | 9
  Unspecified Hearing Loss | 1 | 1
Statistical Analysis 1: Comparison: As-Treated No Growth Hormone vs As-Treated Growth Hormone; Comparison of proportion of patients with any category of hearing loss between As-Treated Growth Hormone group and As-Treated No Growth Hormone; Test type: Superiority or Other; p > 0.999, Fisher Exact

9. Secondary Outcome: Fasting Glucose, Change From Baseline
Description: Change from core study baseline to addendum 2 maximum.
Time Frame: At core study baseline, and at end of 4-year addendum
Population: Patients who were followed for at least 4 years without growth hormone treatment or who received growth hormone for at least 4 years, and who were treated as randomized and had core study baseline and addendum glucose metabolism data.
Measure: Least Squares Mean (Standard Error); unit: mg / dL
Groups:
- Treated-As-Randomized Control: Patients in As-Randomized Control group who at each observed time point remained untreated with growth hormone.
- Treated-As-Randomized Humatrope: Patients in As-Randomized Humatrope group who received Humatrope treatment
Arm/Group | Treated-As-Randomized Control | Treated-As-Randomized Humatrope
Number analyzed (Participants) | 20 | 36
mg / dL | 5.495 (2.455) | 3.003 (1.830)
Statistical Analysis 1: Comparison: Treated-As-Randomized Control vs Treated-As-Randomized Humatrope; Test type: Superiority or Other; p = 0.419, ANOVA; Mean Difference (Final Values) = -2.492, 95% CI [-8.631 to 3.646] — Direction of estimated treatment effect is Humatrope minus Control

10. Secondary Outcome: Maximum Fasting Glucose Value
Description: Maximum measured value over addendum. In special cases an additional measurement is taken at 2 years.
Time Frame: At start and through end of 4-year addendum (up to an additional 2 years)
Population: Patients with addendum data who were followed for at least 4 years without growth hormone treatment (and never received growth hormone) or who received growth hormone for at least 4 years.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | As-Treated No Growth Hormone | As-Treated Growth Hormone
Number analyzed (Participants) | 21 | 39
milligrams per deciliter (mg/dL) | 85.2 (6.6) | 85.2 (10.4)

11. Secondary Outcome: Number of Participants With Any Abnormal Fasting Glucose Value
Description: Indicates if patient had any measured value exceeding threshold of normality at any visit during addendum. Abnormal Fasting Glucose=Fasting Glucose >=100 milligrams per deciliter (mg/dL).
Time Frame: At start and through end of 4-year addendum
Population: Patients with any Addendum 2 glucose metabolism data
Measure: Number; unit: participants
Arm/Group | As-Treated No Growth Hormone | As-Treated Growth Humatrope
Number analyzed (Participants) | 21 | 39
participants | 0 | 3
Statistical Analysis 1: Comparison: As-Treated No Growth Hormone vs As-Treated Growth Humatrope; Test type: Superiority or Other; p = 0.545, Fisher Exact

12. Secondary Outcome: Maximum Fasting Insulin Values
Description: Maximum measured value over addendum. In special cases an additional measurement is taken at 2 years.
Time Frame: At start and through end of 4-year addendum (up to an additional 2 years)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: micro International Units per milliliter
Arm/Group | As-Treated No Growth Hormone | As-Treated Growth Hormone
Number analyzed (Participants) | 21 | 40
micro International Units per milliliter | 9.5 (10.8) | 9.7 (9.3)

13. Secondary Outcome: Number of Participants With Any Abnormal Fasting Insulin Value
Description: Indicates if patient had any measured value exceeding threshold of normality at any visit during addendum. Abnormal Fasting Insulin = Fasting Insulin >=35 micro International Units per milliliter (uIU/mL).
Time Frame: At start and through end of 4-year addendum
Population: Patients with any Addendum 2 glucose metabolism data
Measure: Number; unit: participants
Arm/Group | As-Treated No Growth Hormone | As-Treated Growth Humatrope
Number analyzed (Participants) | 21 | 40
participants | 1 | 2
Statistical Analysis 1: Comparison: As-Treated No Growth Hormone vs As-Treated Growth Humatrope; Test type: Superiority or Other; p > 0.999, Fisher Exact

14. Secondary Outcome: Minimum Fasting Glucose/Insulin Ratio Values
Description: Minimum measured value over addendum. In special cases an additional measurement is taken at 2 years.
Time Frame: At start and through end of 4-year addendum (up to an additional 2 years)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: milligrams per 10^-4 Units (mg/[10^-4]U)
Arm/Group | As-Treated No Growth Hormone | As-Treated Growth Hormone
Number analyzed (Participants) | 21 | 38
milligrams per 10^-4 Units (mg/[10^-4]U) | 12.5 (6.0) | 12.2 (5.3)

15. Secondary Outcome: Number of Participants With Any Abnormal Fasting Glucose/Insulin Ratio Value
Description: Indicates if patient had any measured value below threshold of normality at any visit during addendum. Abnormal Fasting Glucose/Insulin Ratio = Fasting Glucose/Insulin Ratio <=4.5 milligrams per 10^-4 Units (mg/10^-4U).
Time Frame: At start and through end of 4-year addendum
Population: Patients with any Addendum 2 glucose metabolism data. Calculated only for patients with fasting blood <100 mg/dL.
Measure: Number; unit: participants
Arm/Group | As-Treated No Growth Hormone | As-Treated Growth Hormone
Number analyzed (Participants) | 21 | 38
participants | 1 | 3
Statistical Analysis 1: Comparison: As-Treated No Growth Hormone vs As-Treated Growth Hormone; Test type: Superiority or Other; p > 0.999, Fisher Exact

16. Secondary Outcome: Glycosylated Hemoglobin, Change From Baseline
Description: Change from core study baseline to addendum 2 maximum.
Time Frame: At core study baseline, and at end of 4-year addendum
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: percent (%)
Groups:
- Treated-As-Randomized Humatrope: Patients in the As-Randomized Humatrope group who received Humatrope
Arm/Group | Treated-As-Randomized Control | Treated-As-Randomized Humatrope
Number analyzed (Participants) | 20 | 36
percent (%) | 0.215 (0.077) | 0.208 (0.057)
Statistical Analysis 1: Comparison: Treated-As-Randomized Control vs Treated-As-Randomized Humatrope; Test type: Superiority or Other; p = 0.945, ANOVA; Mean Difference (Final Values) = -0.007, 95% CI [-0.199 to 0.186] — Direction of estimated treatment effect is Humatrope minus Control

17. Secondary Outcome: Maximum Glycosylated Hemoglobin
Description: Maximum measured value over addendum. In special cases an additional measurement is taken at 2 years.
Time Frame: At start and through end of 4-year addendum (up to an additional 2 years)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percent (%)
Arm/Group | As-Treated No Growth Hormone | As-Treated Growth Hormone
Number analyzed (Participants) | 21 | 40
percent (%) | 5.0 (0.5) | 5.0 (0.4)

18. Secondary Outcome: Number of Participants With Any Abnormal Glycosylated Hemoglobin (HbA1c) Value
Description: Indicates if patient had any measured value exceeding threshold of normality at any visit during addendum. Abnormal Glycosylated Hemoglobin = HbA1c ≥6.8% (up until 11-May-1998); and then HbA1c ≥6.1% (from 19-May-1998 onwards).
Time Frame: At start and through end of 4-year addendum
Population: Patients with any Addendum 2 glucose metabolism data.
Measure: Number; unit: participants
Arm/Group | As-Treated No Growth Hormone | As-Treated Growth Hormone
Number analyzed (Participants) | 21 | 40
participants | 0 | 0
Statistical Analysis 1: Comparison: As-Treated No Growth Hormone vs As-Treated Growth Hormone; Test type: Superiority or Other; Fisher Exact — P-value cannot be computed since no patients had abnormal result in either comparison group

ADVERSE EVENTS:
Groups:
- Treated-As-Randomized Control: Patients in the As-Randomized Control group who at each observed time point remained untreated with growth hormone.
Arm/Group | Treated-As-Randomized Control | Treated-As-Randomized Humatrope
Serious Adverse Events (participants affected / at risk) | 10/54 | 22/74
Other Adverse Events (participants affected / at risk) | 53/54 | 74/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treated-As-Randomized Control (N=54) | Treated-As-Randomized Humatrope (N=74)
Anemia iron deficiency (Blood and lymphatic system disorders) | 0 | 1
Hypochromic microcytic anemia (Blood and lymphatic system disorders) | 0 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cellulitis of foot (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Stomach flu (Infections and infestations) | 0 | 1
Viral meningitis (Infections and infestations) | 0 | 1
Arm fracture (Injury, poisoning and procedural complications) | 0 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Colonoscopy (Investigations) | 0 | 1
Cystoscopy (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Adenoidectomy (Surgical and medical procedures) | 0 | 1
Aorta coarctation repair (Surgical and medical procedures) | 0 | 1
Appendectomy (Surgical and medical procedures) | 2 | 0
Chest wall repair (Surgical and medical procedures) | 1 | 0
Cholesteatoma removal (Surgical and medical procedures) | 0 | 1
Dental surgery NOS (Surgical and medical procedures) | 0 | 1
Eye muscle operation (Surgical and medical procedures) | 0 | 1
Heart valve operation (Surgical and medical procedures) | 0 | 1
Mastoid operation (Surgical and medical procedures) | 0 | 1
Mastoidectomy (Surgical and medical procedures) | 0 | 1
Orchiectomy (Surgical and medical procedures) | 0 | 1
Pterygium operation (Surgical and medical procedures) | 1 | 1
Scar removal (Surgical and medical procedures) | 1 | 0
Surgical procedure (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0
Tympanoplasty (Surgical and medical procedures) | 0 | 3
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treated-As-Randomized Control (N=54) | Treated-As-Randomized Humatrope (N=74)
Ear ache (Ear and labyrinth disorders) | 6 | 10
Ear discharge (Ear and labyrinth disorders) | 0 | 4
Ear pain (Ear and labyrinth disorders) | 3 | 14
Earache (Ear and labyrinth disorders) | 5 | 8
Hearing loss (Ear and labyrinth disorders) | 2 | 7
Sensorineural hearing loss (Ear and labyrinth disorders) | 3 | 0
Tympanosclerosis (Ear and labyrinth disorders) | 3 | 0
Hypothyroidism (Endocrine disorders) | 7 | 13
Conjunctivitis (Eye disorders) | 2 | 4
Myopia (Eye disorders) | 3 | 4
Abdominal pain (Gastrointestinal disorders) | 9 | 9
Ache stomach (Gastrointestinal disorders) | 0 | 4
Diarrhea (Gastrointestinal disorders) | 11 | 12
Nausea (Gastrointestinal disorders) | 5 | 13
Stomach ache (Gastrointestinal disorders) | 7 | 7
Stomach cramps (Gastrointestinal disorders) | 4 | 4
Stomach pain (Gastrointestinal disorders) | 2 | 6
Upset stomach (Gastrointestinal disorders) | 3 | 5
Vomiting (Gastrointestinal disorders) | 21 | 29
Chest pain (General disorders) | 4 | 1
Fatigue (General disorders) | 4 | 1
Fever (General disorders) | 20 | 36
Pain (General disorders) | 0 | 4
Hay fever (Immune system disorders) | 1 | 7
Multiple allergies (Immune system disorders) | 1 | 6
Bladder infection (Infections and infestations) | 3 | 4
Bronchitis (Infections and infestations) | 5 | 7
Chest cold (Infections and infestations) | 0 | 7
Chickenpox (Infections and infestations) | 5 | 8
Cold (Infections and infestations) | 39 | 42
Cold symptoms (Infections and infestations) | 4 | 7
Common cold (Infections and infestations) | 4 | 5
Ear infection (Infections and infestations) | 12 | 27
Eye infection (Infections and infestations) | 3 | 9
Flu (Infections and infestations) | 20 | 36
Flu syndrome (Infections and infestations) | 6 | 15
Gastroenteritis (Infections and infestations) | 2 | 6
Head cold (Infections and infestations) | 9 | 18
Impetigo (Infections and infestations) | 4 | 6
Otitis externa (Infections and infestations) | 6 | 13
Otitis media (Infections and infestations) | 13 | 31
Pharyngitis (Infections and infestations) | 8 | 11
Rhinitis (Infections and infestations) | 11 | 17
Sinus infection (Infections and infestations) | 1 | 5
Sinusitis (Infections and infestations) | 3 | 7
Stomach flu (Infections and infestations) | 6 | 6
Streptococcal sore throat (Infections and infestations) | 4 | 9
Throat infection (Infections and infestations) | 7 | 8
Tonsillitis (Infections and infestations) | 5 | 6
Upper respiratory infection (Infections and infestations) | 14 | 13
Upper respiratory tract infection (Infections and infestations) | 9 | 8
Urinary tract infection (Infections and infestations) | 3 | 5
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 5
Head injury (Injury, poisoning and procedural complications) | 3 | 2
Knee pain (Musculoskeletal and connective tissue disorders) | 1 | 8
Leg pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Low back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Osteopenia (Musculoskeletal and connective tissue disorders) | 4 | 2
Scoliosis (Musculoskeletal and connective tissue disorders) | 8 | 6
Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Dizziness (Nervous system disorders) | 4 | 7
Headache (Nervous system disorders) | 25 | 46
Intermittent headache (Nervous system disorders) | 3 | 12
Depression (Psychiatric disorders) | 4 | 6
Cramps menstrual (Reproductive system and breast disorders) | 2 | 4
Dysmenorrhea (Reproductive system and breast disorders) | 2 | 4
Menstrual cramps (Reproductive system and breast disorders) | 7 | 7
Primary ovarian failure (Reproductive system and breast disorders) | 4 | 5
Spotting vaginal (Reproductive system and breast disorders) | 4 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Congestion nasal (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 27
Coughing (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 17
Nasal discharge (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Sore throat (Respiratory, thoracic and mediastinal disorders) | 28 | 37
Throat sore (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 8
Eczema (Skin and subcutaneous tissue disorders) | 4 | 4
Ingrown toe nail (Skin and subcutaneous tissue disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 8 | 8
Dental surgery NOS (Surgical and medical procedures) | 1 | 4
Dental treatment (Surgical and medical procedures) | 8 | 6
Ear tube insertion (Surgical and medical procedures) | 1 | 4
Mole excision (Surgical and medical procedures) | 2 | 5
Myringotomy (Surgical and medical procedures) | 1 | 8
Tooth extraction (Surgical and medical procedures) | 3 | 3
Tympanoplasty (Surgical and medical procedures) | 0 | 4
Aortic dilatation (Vascular disorders) | 3 | 1
Blood pressure high (Vascular disorders) | 3 | 1
Hypertension (Vascular disorders) | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days